CLINICAL TRIAL: NCT05561205
Title: Repetitive Transcranial Magnetic Stimulation for Apathy Clinical Trial (REACT)
Brief Title: rTMS for Apathy Clinical Trial
Acronym: REACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUN-5342
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Apathy in Dementia; Dementia; Mild Behavioural Impairment; Mild Cognitive Impairment; Neurocognitive Disorders
Keywords: Apathy; Alzheimer's disease; Neurocognitive disorder; Mild behavioural impairment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Neurocognitive Disorders; Lethargy | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS + methylphenidate (Experimental): repetitive transcranial magnetic stimulation (rTMS) and methylphenidate
  Interventions: Device: rTMS; Drug: methylphenidate
- rTMS only (Experimental): repetitive transcranial magnetic stimulation (rTMS) only
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — repetitive transcranial magnetic stimulation
Drug: methylphenidate — methylphenidate
  Arms: rTMS + methylphenidate

SUMMARY:
Apathy is a common, early, and disabling symptom in dementias and mild behavioural impairment such as Alzheimer's disease (AD) and is characterized by lack of interest and enthusiasm. Both repetitive transcranial magnetic stimulation (rTMS), a form of non-invasive brain stimulation, and methylphenidate, a medication, have been shown to improve apathy. This pilot study will investigate rTMS as a treatment for apathy in neurocognitive disorders and mild behavioural impairment in individuals receiving methylphenidate and individuals not receiving medication for apathy.

ELIGIBILITY:
Inclusion Criteria:

* mild or major neurocognitive disorder OR mild behavioural impairment
* Apathy for at least 4 weeks
* Stable dose of medication (>4 weeks) that may affect cognition or behaviour
* Care partner who spends at least 10 hours a week with the subject

Exclusion Criteria:

* Current major depressive episode
* Agitation, delusions, hallucination
* Medical contraindications to rTMS
* Currently taking an amphetamine product
* Central nervous system abnormalities, Tourette's syndrome, or motor tics
* Current participation in another clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory-apathy | 2 weeks
  Measure of apathy on a scale from 0 to 12 with a higher score indicating greater apathy

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada